CLINICAL TRIAL: NCT00014443
Title: A Pilot Study Of Hycamtin (Topotecan) And Thalomid (Thalidomide) In Patients With Recurrent Malignant Gliomas
Brief Title: Topotecan and Thalidomide in Treating Patients With Recurrent or Refractory Malignant Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068544; RUSH-G101; NCI-V01-1651
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — Thalidomide; Topotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: thalidomide
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of combining topotecan and thalidomide in treating patients who have recurrent or refractory malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine tumor response rate, duration of response, time to disease progression, and overall survival of patients with recurrent or refractory malignant glioma treated with topotecan and thalidomide.
* Determine safety and tolerance of this regimen in these patients.

OUTLINE: Patients receive topotecan IV continuously on days 1-21 and oral thalidomide daily on days 1-28. Treatment repeats every 28 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or progressive supratentorial glioblastoma or anaplastic astrocytoma
* Measurable disease by MRI or CT scan
* No gliomatosis cerebri, anaplastic oligodendroglioma, or anaplastic oligoastrocytoma
* Concurrent registration for the System for Thalidomide Education and Prescribing Safety (S.T.E.P.S.) program

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL

Renal:

* Creatinine less than 1.6 mg/dL

Other:

* No other concurrent malignancy except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception 1 month prior to, during, and for 1 month after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 2 prior chemotherapy regimens in adjuvant or metastatic setting
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Concurrent anticonvulsants allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2000-08 (Actual); Primary Completion 2003-08 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pam G. Khosla, MD, Study Chair — Rush University Medical Center
Locations (1):
- Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois, United States